CLINICAL TRIAL: NCT04238156
Title: Hypopressive Abdominal Exercise Effectiveness in Postpartum Abdominal Diastasis, Tone of the Transverse Muscle and the Pelvic Floor Muscles - Case Series
Brief Title: Hypopressive Abdominal Exercise in Postpartum Abdominal Diastasis
Acronym: HipoDiastasi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Córdoba (Other)
Responsible Party: Principal Investigator, Francisco Alburquerque-Sendín, Ph D, Associate Professor, Universidad de Córdoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HipoDiastasis4073-2018
Record Dates: First submitted 2020-01-15; First posted 2020-01-23 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Abdominal Diastasis
Keywords: Postpartum; Hypopressive abdominal exercises; Pelvic floor muscles

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypopressive abdominal exercises (Experimental): Hypopressive abdominal exercises will be performed in basic postures (standing, sitting and supine position). In each posture, three slow cost-diaphragmatic respiration will be performed followed by an expiratory apnea and a rib cage opening, during 2 to 10 seconds, and an exhalation of 10 to 30 seconds. Each exercise will be repeated three times.
  There will be 3 stages of application throughout the 12 intervention sessions, supervised by a physical therapist:
  First stage: To explain the concept of hypopressive respiration and how to perform it.
  Second stage: To explain and apply the hypopressive abdominal exercises: 1. Axial auto-elongation (reducing curvatures in the sagittal plane); 2. Cervical auto-elongation (chin toward the neck); 3. Moving forward of gravity axis; 4. Activation of the shoulder girdle (shoulder joint decoaptation); 5. Slight knee flexion; 6. Dorsal ankle flexion.
  Third stage: To review and update all the exercises, increasing their intensity.
  Interventions: Other: Hypopressive abdominal exercises

INTERVENTIONS:
Other: Hypopressive abdominal exercises — Three sessions per week during four consecutive weeks (Total: 12 sessions). Each session time: 30 minutes.

SUMMARY:
The prevalence of abdominal diastasis is high in postpartum. The abdominal diastasis can impair the body posture, the of lumbo-pelvic stability and movement, or breathing. Exercises focused on the transversus abdominis muscle have been proposed as a therapeutic approach for abdominal diastasis.

Hypopressive abdominal exercises have been used for postpartum recovery, for specific pathologies related to pregnancy (low back pain, pelvic floor dysfunction ...) and even for the rehabilitation of spinal pathologies. However, there is a lack of studies that determine its effectiveness and clinical utility.

The aim of the study will be to analyze the effects of Hypopressive abdominal exercises on postpartum abdominal diastasis, the tone of the transverse abdominal muscle and the pelvic floor musculature.

A case series design will be applied, with weekly assessment of the outcomes after the intervention and two months after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* primiparous or multiparous
* abdominal diastasis previously diagnosed
* commitment to perform, at least, 80% of the exercises
* signed informed consent

Exclusion Criteria:

* BMI > 40 Kg/m2
* pelvic floor disorders before childbirth
* drugs with effects on continence or functional properties of the pelvic floor muscles
* treatment for abdominal diastasis in the last 6 months
* systemic disease that impairs pelvic floor physiology and urination
* menopause
* contraindications to the practice of physical exercise and physical therapy

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
Abdominal Diastasis - Baseline | Pre-intervention
  Supraumbilical distance between the rectus abdominis
  * Assessment tool: caliper (electronic, calibrated, precision: 1 mm)
  * Subject position: supine
  * Localization: 3 cm, 6 cm, 9 cm, 12 cm supraumbilical
Abdominal Diastasis - post-intervention 1 | Immediately after the intervention
  Supraumbilical distance between the rectus abdominis
  * Assessment tool: caliper (electronic, calibrated, precision: 1 mm)
  * Subject position: supine
  * Localization: 3 cm, 6 cm, 9 cm, 12 cm supraumbilical
Abdominal Diastasis - post-intervention 2 | One month after the intervention
  Supraumbilical distance between the rectus abdominis
  * Assessment tool: caliper (electronic, calibrated, precision: 1 mm)
  * Subject position: supine
  * Localization: 3 cm, 6 cm, 9 cm, 12 cm supraumbilical
Abdominal Diastasis - post-intervention 3 | Two months after the intervention
  Supraumbilical distance between the rectus abdominis
  * Assessment tool: caliper (electronic, calibrated, precision: 1 mm)
  * Subject position: supine
  * Localization: 3 cm, 6 cm, 9 cm, 12 cm supraumbilical

SECONDARY OUTCOMES:
Abdominal tonometry - Baseline | Pre-intervention
  Tonometric evaluation on the white line (linea alba) and the abdominal muscles
  * Assessment tool: (MyotonPro (R))
  * Subject position: supine
  * Localization: 3 cm, 6 cm, 9 cm, 12 cm supraumbilical
Perineal tonometry - Baseline | Pre-intervention
  Tonometric evaluation on the perineal muscles
  * Assessment tool: (MyotonPro (R))
  * Subject position: supine
  * Localization: 3 cm, 6 cm, 9 cm, 12 cm supraumbilical
Waist circumference - Baseline | Pre-intervention
  Waist circumference
  * Assessment tool: tape measure (flexible, precision: 1mm)
  * Subject position: standing
  * Localization: minimum perimeter
Chest circumference - Baseline | Pre-intervention
  Chest circumference
  * Assessment tool: tape measure (flexible, precision: 1mm)
  * Subject position: standing
  * Localization: maximum perimeter
Abdominal tonometry - post-intervention 1 | Immediately after the intervention
  Tonometric evaluation on the white line (linea alba) and the abdominal muscles
  * Assessment tool: (MyotonPro (R))
  * Subject position: supine
  * Localization: 3 cm, 6 cm, 9 cm, 12 cm supraumbilical
Perineal tonometry - post-intervention 1 | Immediately after the intervention
  Tonometric evaluation on the perineal muscles
  * Assessment tool: (MyotonPro (R))
  * Subject position: supine
  * Localization: 3 cm, 6 cm, 9 cm, 12 cm supraumbilical
Waist circumference - post-intervention 1 | Immediately after the intervention
  Waist circumference
  * Assessment tool: tape measure (flexible, precision: 1mm)
  * Subject position: standing
  * Localization: minimum perimeter
Chest circumference - post-intervention 1 | Immediately after the intervention
  Chest circumference
  * Assessment tool: tape measure (flexible, precision: 1mm)
  * Subject position: standing
  * Localization: maximum perimeter
Abdominal tonometry - post-intervention 2 | One month after the intervention
  Tonometric evaluation on the white line (linea alba) and the abdominal muscles
  * Assessment tool: (MyotonPro (R))
  * Subject position: supine
  * Localization: 3 cm, 6 cm, 9 cm, 12 cm supraumbilical
Perineal tonometry - post-intervention 2 | One month after the intervention
  Tonometric evaluation on the perineal muscles
  * Assessment tool: (MyotonPro (R))
  * Subject position: supine
  * Localization: 3 cm, 6 cm, 9 cm, 12 cm supraumbilical
Waist circumference - post-intervention 2 | One month after the intervention
  Waist circumference
  * Assessment tool: tape measure (flexible, precision: 1mm)
  * Subject position: standing
  * Localization: minimum perimeter
Chest circumference - post-intervention 2 | One month after the intervention
  Chest circumference
  * Assessment tool: tape measure (flexible, precision: 1mm)
  * Subject position: standing
  * Localization: maximum perimeter
Abdominal tonometry - post-intervention 3 | Two months after the intervention
  Tonometric evaluation on the white line (linea alba) and the abdominal muscles
  * Assessment tool: (MyotonPro (R))
  * Subject position: supine
  * Localization: 3 cm, 6 cm, 9 cm, 12 cm supraumbilical
Perineal tonometry - post-intervention 3 | Two months after the intervention
  Tonometric evaluation on the perineal muscles
  * Assessment tool: (MyotonPro (R))
  * Subject position: supine
  * Localization: 3 cm, 6 cm, 9 cm, 12 cm supraumbilical
Waist circumference - post-intervention 3 | Two months after the intervention
  Waist circumference
  * Assessment tool: tape measure (flexible, precision: 1mm)
  * Subject position: standing
  * Localization: minimum perimeter
Chest circumference - post-intervention 3 | Two months after the intervention
  Chest circumference
  * Assessment tool: tape measure (flexible, precision: 1mm)
  * Subject position: standing
  * Localization: maximum perimeter

CONTACTS AND LOCATIONS:
Overall Officials: Daiana Priscila Rodrigues-de-Souza, PhD, Study Director — Universidad de Córdoba; Miriam Ramírez Jiménez, Phys Ther, Principal Investigator — Universidad de Córdoba
Locations (1):
- University of Córdoba, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: No